CLINICAL TRIAL: NCT06711588
Title: Automatic Activity-Dependent and Phase-Varying Prosthetic Foot Stiffness Modulation to Improve Balance Control in Individuals With Lower-Limb Amputations
Brief Title: Automatic Prosthetic Foot Stiffness Modulation to Improve Balance
Acronym: OSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 1817327; 1R01HD111514-01A1 (NIH)
Record Dates: First submitted 2024-11-24; First posted 2024-12-02 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Lower Limb Amputation Below Knee
Keywords: lower limb prosthesis; transtibial amputation; below knee amputation; biomechanics; gait

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (9):
- Walking on 0% slope at self-selected speed (Experimental): All participants will walk on a treadmill, in a straight line, on a 0% slope, at their self-selected walking speed determined while walking overground.
  Interventions: Device: As-prescribed stiffness; Device: Two categories stiffer than the as-prescribed stiffness; Device: Two categories less stiff than the as-prescribed stiffness
- Walking on 0% slope at 15% slower than self-selected speed (Experimental): All participants will walk on a treadmill, in a straight line, on a 0% slope, at a speed that is 15% slower than their self-selected walking speed determined while walking overground.
  Interventions: Device: As-prescribed stiffness; Device: Two categories stiffer than the as-prescribed stiffness; Device: Two categories less stiff than the as-prescribed stiffness
- Walking on 0% slope at 15% faster than self-selected speed (Experimental): All participants will walk on a treadmill, in a straight line, on a 0% slope, at a speed that is 15% faster than their self-selected walking speed determined while walking overground.
  Interventions: Device: As-prescribed stiffness; Device: Two categories stiffer than the as-prescribed stiffness; Device: Two categories less stiff than the as-prescribed stiffness
- Walking up an 8% slope at self-selected speed (Experimental): All participants will walk on a treadmill, in a straight line, up an 8% slope, at their self-selected walking speed determined while walking overground up an 8% slope.
  Interventions: Device: As-prescribed stiffness; Device: Two categories stiffer than the as-prescribed stiffness; Device: Two categories less stiff than the as-prescribed stiffness
- Walking down an 8% slope at self-selected speed (Experimental): All participants will walk on a treadmill, in a straight line, down an 8% slope, at their self-selected walking speed determined while walking overground up an 8% slope.
  Interventions: Device: As-prescribed stiffness; Device: Two categories stiffer than the as-prescribed stiffness; Device: Two categories less stiff than the as-prescribed stiffness
- Walking on 0% slope at self-selected speed while hand carrying a 5 kg load on their prosthetic side (Experimental): All participants will walk on a treadmill, in a straight line, on a 0% slope, at their self-selected walking speed determined while walking overground, while carrying a 5 kg load in one hand on their prosthetic side.
  Interventions: Device: As-prescribed stiffness; Device: Two categories stiffer than the as-prescribed stiffness; Device: Two categories less stiff than the as-prescribed stiffness
- Walking on uneven terrain at self-selected speed (Experimental): All participants will walk on an uneven terrain treadmill, in a straight line, on a 0% slope, at their self-selected walking speed determined while walking on the uneven terrain treadmill.
  Interventions: Device: As-prescribed stiffness; Device: Two categories stiffer than the as-prescribed stiffness; Device: Two categories less stiff than the as-prescribed stiffness
- Walking around a 2-meter diameter circle with the prosthesis on the inside of the circle (Experimental): All participants will walk overground while following the outline of a 2-meter diameter circle, at their self-selected walking speed determined while walking around the circle, with their prosthetic limb on the inside of the circle.
  Interventions: Device: As-prescribed stiffness; Device: Two categories stiffer than the as-prescribed stiffness; Device: Two categories less stiff than the as-prescribed stiffness
- Walking around a 2-meter diameter circle with the prosthesis on the outside of the circle (Experimental): All participants will walk overground while following the outline of a 2-meter diameter circle, at their self-selected walking speed determined while walking around the circle, with their prosthetic limb on the outside of the circle.
  Interventions: Device: As-prescribed stiffness; Device: Two categories stiffer than the as-prescribed stiffness; Device: Two categories less stiff than the as-prescribed stiffness

INTERVENTIONS:
Device: As-prescribed stiffness — A novel prosthesis that includes a low-profile prosthetic foot whose stiffness category is determined by the person's body weight and activity level (standard clinical practice).
Device: Two categories stiffer than the as-prescribed stiffness — A novel prosthesis that includes a low-profile prosthetic foot whose stiffness category is two categories stiffer than the as-prescribed stiffness.
Device: Two categories less stiff than the as-prescribed stiffness — A novel prosthesis that includes a low-profile prosthetic foot whose stiffness category is two categories less stiff than the as-prescribed stiffness.

SUMMARY:
The goal of this clinical trial is to identify prosthesis stiffness that optimizes balance control in individuals with below knee amputations. The main question this clinical trial will answer is:

• Is there an optimal stiffness that improves balance control for specific ambulatory activities and users? Participants will wear a novel prosthesis assembled with three prosthetic feet with a range of stiffness levels: each individual's clinically-prescribed foot stiffness and ± two stiffness categories. While wearing the study prostheses, participants will perform nine ambulatory activities of daily living (walking at different speeds, turning, ramp ascent/descent, while carrying a load, and while walking on uneven terrain).

DETAILED DESCRIPTION:
Individuals with lower limb amputations are at higher risk of falling compared to able-bodied and other clinical populations and are more likely to sustain life-altering injuries. The higher fall risk is primarily due to the loss of the muscles crossing the ankle, which are critical to maintaining balance control. Prosthetic devices are designed to provide appropriate stiffness for needed stability and support. While research has shown the optimal stiffness to maintain balance varies across ambulatory activities (e.g., straight walking versus turning), most clinically prescribed prosthetic devices are passive and only provide a fixed stiffness level. The one commercially available, powered prosthetic ankle-foot has not been shown to restore balance control. Thus, a prosthetic device that actively adjusts ankle stiffness across different ambulatory activities is critically needed to advance the field and improve balance control for those with lower-limb amputations. The goal of this clinical trial is to identify prosthesis stiffness that optimizes balance control in individuals with below knee amputations as they perform typical ambulatory activities of daily living. By matching the ankle stiffness to the task requirements, we believe we will significantly improve balance control and decrease fall risk for those with lower-limb amputations.

Each participant will be fit with a novel prosthesis that includes a low-profile prosthetic foot whose stiffness category will be determined by their body weight and activity level (standard clinical practice), a prosthetic foot whose stiffness category is two categories stiffer, and another whose stiffness is two categories less stiff. Participants will continue to use their existing prosthetic socket and suspension system, but their pylon length will be adjusted as needed. While wearing the different study prostheses in randomized order, nine ambulatory activities will be performed motion capture laboratory.

1. Walking on level ground at self-selected speed.
2. Walking on level ground at 15% slower than self-selected speed.
3. Walking on level ground at 15% faster than self-selected speed.
4. Walking up an 8% slope at self-selected speed.
5. Walking down an 8% slope at self-selected speed.
6. Walking on level ground at self-selected speed while carrying a 5 kg load in one hand on their prosthetic side.
7. Walking on level but uneven terrain at self-selected speed.
8. Walking a 2-meter diameter circle at self-selected speed with the prosthetic side on the inside of the circle.
9. Walking a 2-meter diameter circle at self-selected speed with the prosthetic side on the outside of the circle.

Ambulatory activities 1 through 6 will be performed on an instrumented treadmill. The load to be carried in activity 6 will be configured as a grocery bag with handles. Activity 7 will be performed on a rocky terrain treadmill. Activities 8 and 9 will be performed overground across five force plates embedded in the laboratory floor while following the outline of a 2-meter diameter circle. Rest breaks during all activities will be provided as needed.

The data from these experiments will be used to calculate the peak-to-peak range of the frontal plane whole-body angular momentum (a measure of balance control). We hypothesize that an optimal user-specific stiffness profile exists that maximizes balance control (i.e., minimizes the peak-to-peak range of frontal plane whole-body angular momentum over the gait cycle) for each ambulatory activity.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial (below-knee) amputation
* Been fit with a prosthesis and used it for at least 6 months
* Wear the prosthesis for 4 or more hours on average per day
* Be at least one-year post-amputation
* Able to walk on a treadmill

Exclusion Criteria:

* Presence of disorder, pain, or injury other than amputation that interferes with gait
* Current skin irritation or injury on residual limb
* Use of an assistive device for walking (cane, walker, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Peak-to-peak range of the frontal plane whole-body angular momentum | During study visit (approximately 3 hours)
  Frontal plane whole-body angular momentum is a measure of the extent to which a person will rotate in the frontal plane in the absence of an external force or torque. The peak-to-peak range quantifies how much this metric varies and is used to describe a person's balance.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Klute, PhD, Principal Investigator — US Department of Veterans Affairs; Richard Neptune, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- VA Puget Sound Healthcare System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data sets of all IPD collected throughout the trial will be made available, in machine-readable format, on the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub (DASH). The de-identification procedures will follow 164.514(a) of the HIPAA Privacy Rule.
Supporting Information: Study Protocol, ICF
Time Frame: Publication-associated datasets will be submitted to DASH at least 4 months prior to publication so that data can be shared on or before the initial publication date. The full study dataset will be submitted to DASH at least 6 months prior to the end of the award period. DASH does not currently have any data deprecation or sunsetting protocols, allowing shared data to be preserved for the foreseeable future.
Access Criteria: DASH is an NIH controlled-access data repository. The NICHD DASH Data Access Committee reviews all requests to access DASH data from identity-verified requesters to determine whether the proposed use is scientifically and ethically appropriate and does not conflict with constraints or research data use limitations identified by the institutions that submitted the research data. The Recipient's institution and the Recipient must sign and agree to the terms and conditions in the NICHD DASH Data Use Agreement for accessing research data.